CLINICAL TRIAL: NCT06815874
Title: Recurrence of Thromboembolic Venous Disease of Atypical Location
Brief Title: Recurrence of Thromboembolic Venous Disease of Atypical Location (RUSE)
Acronym: RUSE
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0345 - RUSE
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-11

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
RUSE is a retrospective data-based study designed to assess the frequency, characteristics and phenotype of documented recurrences of thromboembolic venous disease in atypical locations.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18,
* Affiliated to "sécurité sociale"
* Having at least one episode of atypical localisation of VTE at Brest University Hospital

Exclusion Criteria:

* Patients under legal protection
* Minors
* Refusal to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient with documented atypical localisation of VTE
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Documented recurrence after previous VTE in atypical localisations | 01/01/2005 to 01/11/2024
  All forms of VTE of typical (DVT and PE) and atypical location, muscular venous thrombosis and documented superficial venous thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement